CLINICAL TRIAL: NCT06152692
Title: Circadian Intraocular Pressure Patterns in Patients With Sleep Apnea Syndrome and Treatment With Continuous Air Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Principal Investigator, Ferran Barbe, Chair Respiratory Medicine, Sociedad Española de Neumología y Cirugía Torácica
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: PI15/02179
Record Dates: First submitted 2023-11-21; First posted 2023-12-01 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Circadian rhythms; Intraocular pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OSA + CPAP (Experimental): OSA + CPAP
  Interventions: Device: Continuous positive airway pressure
- OSA + sham CPAP (Placebo Comparator): OSA + sham CPAP
  Interventions: Device: SHAM Continuous positive airway pressure
- Control (No Intervention): Control

INTERVENTIONS:
Device: SHAM Continuous positive airway pressure — Placebo treatment
  Other Names: SHAM CPAP
  Arms: OSA + sham CPAP
Device: Continuous positive airway pressure — Continuous positive airway pressure treatment for patients randomized to CPAP treatment group
  Other Names: CPAP
  Arms: OSA + CPAP

SUMMARY:
The purpose of this study is to evaluate the influence of sleep apnea-hypopnea syndrome (SAHS) syndrome and treatment with continuous air pressure (CPAP) on the circadian intraocular pressure (IOP) patterns and its structural impact on the nerve fiber layer of the retina to analize the relationship between SAHS and glaucoma.

OBJECTIVES: 1. To study the PIO and its fluctuations in patients with SAHS before starting treatment with CPAP. Objective 2. To assess the effect of CPAP on circadian IOP patterns. 3. Evaluate the effect of changes in IOP in patients with OSA treated with CPAP in the nerve fiber layer of the retina.

METHODS: A prospective study to be monitored continuously for 24 hours IOP by contact lens device Sensimed Triggerfish (Sensimed AG, Switzerland). Objective 1. To monitore and compare the IOP for 24 hours at 74 patients diagnosed with SAHS before starting treatment with CPAP and 37 patients without OSA. Objective 2. To study the impact of CPAP treatment by a study design in two stages CPAP / sham CPAP. A first monitoring of IOP will be compared before starting treatment with CPAP, with monitoring a month (CPAP-sham CPAP) and 12 months after initiation of treatment with CPAP. Objective 3. To correlate the values obtained from the monitoring of IOP in the thickness of the nerve fiber layer of the retina, as measured by optical coherence tomography, at baseline and at 12 months after starting treatment with CPAP.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age
* Seeking a sleep study using a cardio-respiratory polygraph study
* Having spherical refraction between -5D and 3D, cylinder correction <2D, as well as a slit lamp examination with anterior chamber normal and an open irido-corneal angle

Exclusion Criteria:

* Presence of severe drowsiness or risk profession that requires urgent treatment with CPAP
* Any known intolerance to silicone, any alteration in the anterior pole of the eye that contraindicates the use of a contact lens, severe dry eye, keratoconus or any other corneal alteration, a history of conventional intraocular or laser surgery, whether for cataracts, glaucoma, refractive or retina surgery.
* Glaucoma patients will be excluded at the start of the study.
* When both eyes of each patient meet the inclusion criteria, the investigator will randomly select the eye to be studied.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2016-01; Primary Completion 2018-06 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Circadian rhythms | At baseline and 12 months
  Compare the circadian rhythms of continuously measured intraocular pressure for 24 hours between patients diagnosed with OSA before initiating CPAP treatment and a group of subjects without OSA.
Circadian intraocular pressure patterns | At baseline, 1 month and 12 months
  Evaluate the effect of CPAP on circadian intraocular pressure patterns after one month and 12 months after starting OSA treatment with CPAP.
IOP-followed patterns | At baseline and 12 months
  Correlate IOP-followed patterns for 24 hours in OSA patients with changes in retinal nerve fiber layer thickness from the start of the study and after 12 months of follow-up.

SECONDARY OUTCOMES:
Circadian rhythms | At baseline and 12 months
  Correlate circadian rhythms followed by IOP as well as changes in the retinal nerve fiber layer with cardio-respiratory polygraphic variables to detect possible risk factors for glaucoma among the OSA population.
OSA and lax eyelid syndrome (SPL) | At baseline and 12 months
  Analyze whether OSA patients who also have lax eyelid syndrome (SPL) have higher or more fluctuating intraocular pressure values that help explain the higher prevalence of glaucoma among patients with OSA and SPL.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Arnau de Vilanova, Lleida, Spain